CLINICAL TRIAL: NCT06544447
Title: Transcutaneous Auricular Vagus Nerve Stimulation in Dry Eye Disease With Meibomian Gland Dysfunction, A Randomized Clinical Trial
Brief Title: Transcutaneous Auricular Vagus Nerve Stimulation in Dry Eye Disease With Meibomian Gland Dysfunction
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Beijing Tongren Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: taVNS-DE-2024
Record Dates: First submitted 2024-08-06; First posted 2024-08-09 (Actual); Last update posted 2024-08-09 (Actual); Status verified 2024-08

CONDITIONS: Dry Eye
Keywords: Dry eye,
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Intervention Model Description: Dry Eye Disease With Meibomian Gland Dysfunction
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- taVNS group (Experimental)
  Interventions: Device: taVNS; Drug: Hyaluronic acid eye drops
- Control Group (Sham Comparator)
  Interventions: Device: taVNS; Drug: Hyaluronic acid eye drops

INTERVENTIONS:
Device: taVNS — taVNS device (Elmmedicare, EC100, Shenzhen, China) was used to apply stimulation for patients. Stimulation parameters comprised an electrical current of 1 mA at a frequency of 20 Hz, with a waveform width of 1 ms. Repurposed off-the-shelf devices were utilized for this purpose, with the stimulator generating single square-wave pulses lasting 1 ms each. Enhancing conductivity was achieved by wiping the ear with tap water.
  The electrodes were placed on the cymba conchae and concha around the affected ear, which is the region of rich vagus nerve branch distribution. Patients in control group were applied using the same stimulator, stimulation parameters and same sessions. However, the electrodes were placed on the antihelix around the affected ear, which is the region of few vagus nerve branch distribution.
Drug: Hyaluronic acid eye drops — Participants in both groups received hyaluronic acid eye drops (HYLO COMOD® eye drops, Ursapharm, Ltd., Germany) with the treatment of 3 times a day.

SUMMARY:
Objective: To evaluate the effect of transcutaneous auricular vagus nerve stimulation (taVNS) for the patients with dry eye disease with meibomian gland dysfunction.

Methods: We enrolled 270 patients at Beijing Tongren Hospital. All treatments were self-administered by the patients at home after training at the hospital. Patients completed questionnaires at baseline, 1 month, 3 months, and 6 months.

OSDI score, TBUT, OPAS, NPSI-eye, and Schirmer I expressibility and secretion score to evaluate the therapeutic effects. A difference of P < 0.05 was considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

1. Age >=18 and Age <=65.
2. Clinical diagnosis of dry eye disease with meibomian gland dysfunction.

Exclusion Criteria:

1. History of depression, tumors, thyroid disease, diabetes, cardiac diseases.
2. History of Otorhinolaryngology surgery.
3. Pregnant or lactating women.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 135 (Estimated)
Dates: Start 2021-06-01 (Actual); Primary Completion 2024-10-01 (Estimated); Study Completion 2024-10-01 (Estimated)

PRIMARY OUTCOMES:
OSDI | Baseline, month 1, 3, and 6
  Ocular Surface Disease Index (OSDI) questionnaire: The OSDI questionnaire is designed to assess the severity of symptoms and the impact of ocular surface diseases, such as dry eye disease, on a patient's quality of life.

SECONDARY OUTCOMES:
OPAS | Baseline, month 1, 3, and 6
  Ocular Surface Disease Index-Personalized Assessment Score (OPAS): The OPAS is a tailored version of the traditional Ocular Surface Disease Index (OSDI). It is designed to offer a more personalized assessment of ocular surface diseases by adapting the standard questionnaire to reflect individual patient experiences and symptoms more accurately. The personalized nature of OPAS aims to offer a more precise measure of how the disease impacts the patient's quality of life and daily functioning.
NPSI-eye | Baseline, month 1, 3, and 6
  Neuropathic Pain Symptom Inventory - Eye (NPSI-eye): The NPSI-eye is a specialized tool designed to assess neuropathic pain symptoms specifically in the context of eye conditions. It helps in identifying and quantifying symptoms associated with neuropathic pain in the ocular region. Higher scores indicate more severe or frequent neuropathic pain symptoms.
TBUT | Baseline, month 1, 3, and 6
  Tear Breakup Time (TBUT): TBUT is a diagnostic test used to evaluate the stability of the tear film and diagnose dry eye disease. It measures the time it takes for dry spots to appear on the corneal surface after blinking while using a fluorescent dye. A shorter TBUT indicates less stable tear film, which is often associated with dry eye disease.
SchirmerI | Baseline, month 1, 3, and 6
  The Schirmer I test assesses tear production to diagnose dry eye syndrome. The length of the wetting is measured in millimeters. A lower measurement indicates reduced tear production, suggesting dry eye disease.

CONTACTS AND LOCATIONS:
Locations (1):
- China Beijing TongRen Hospital, Capital Medical University Beijing, China, Beijing, Beijing Municipality, China